CLINICAL TRIAL: NCT04477551
Title: The Effects of Diode Laser as an Adjunct to Non-surgical Periodontal Treatment on Periodontal Status in Patients With Stage III-IV Periodontitis: a Randomized Controlled Trial
Brief Title: The Effects of Diode Laser as an Adjunct to Non-surgical Periodontal Treatment on Periodontal Status in Patients With Stage III-IV Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Associate Professor Momen Atieh, Chair and Associate Professor (Periodontology), Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBRU/IRB/2020/006
Record Dates: First submitted 2020-07-03; First posted 2020-07-20 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Lasers, Semiconductor; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diode laser (device) with scaling and root planing (Experimental): Diode laser (device) with conventional scaling and root planing
  Interventions: Procedure: Diode laser (device) with scaling and root planing
- Conventional scaling and root planing (Active Comparator): Conventional scaling and root planing
  Interventions: Procedure: Conventional scaling and root planing

INTERVENTIONS:
Procedure: Diode laser (device) with scaling and root planing — Combined use of diode laser device and scaling instruments to remove plaque and calculus from the surface of the roots of teeth.
  Arms: Diode laser (device) with scaling and root planing
Procedure: Conventional scaling and root planing — Use of scaling instruments to remove plaque and calculus from the surface of the roots of teeth.
  Arms: Conventional scaling and root planing

SUMMARY:
Periodontal disease is serious and global chronic disease. The prevalence of periodontal diseases in United Arab Emirates is not clear but data from Dubai Health Authority showed that one in five patients has received periodontal treatment in recent years.

Several studies reported the additional benefits provided by the use of diode laser in combination with ultrasonic debridement in the treatment of gum disease. The use of diode laser may debridement of deep pocketing areas while improving healing of gum tissues.

The aim of the study is to compare the effect of removing bacterial deposit (biofilm) from deep tooth pocket using combined diode laser and conventional pocket debridement versus conventional pocket debridement alone on tooth supporting tissue parameters in patients with advanced gum disease (periodontitis).

Methodology: A total of 22 patients with advanced gum disease will be randomly allocated to two groups: a control group, which will receive conventional pocket debridement and a test group which will receive ultrasonic debridement with diode laser. Gum measurements will be recorded by a masked calibrated examiner at six points for each tooth and patients' postoperative experience and satisfaction will be assessed using special forms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over.
* Diagnosed with unstable generalised periodontitis, stage III-IV and grade B or C.
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion Criteria:

* Received periodontal treatment in the last 12 months.
* Received systemic antibiotic in the last 6 months.
* Pregnancy or lactating participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-10-28 (Estimated); Study Completion 2023-10-28 (Estimated)

PRIMARY OUTCOMES:
Full mouth plaque score (FMPS). | Change from baseline FMPS at six months
  The plaque score is calculated by expressing as a percentage the number of surfaces harbouring plaque related to the total number of tooth surfaces.
Full mouth bleeding score (FMBS). | Change from baseline FMBS at six months
  The bleeding score is calculated by expressing as a percentage the number of sites that bleed upon probing in relation to the total number of tooth sites.
Probing pocket depth (PPD). | Change from baseline PPDs at six months
  PPD is the depth from the free gingival margin to the base of the sulcus and it is measured in millimeters at several locations around the whole circumference of the tooth.
Clinical attachment level (CAL). | Change from baseline CALs at six months
  CAL is calculated from a fixed reference point (cementoenamel junction or CEJ), and it is computed by calculating the distance from the CEJ to the base of the pocket in millimeters.
Number of sites PPDs ≥ 6 mm. | Change from baseline number of sites with PPDs ≥ 6 mm at six months
  Number of sites with PPDs ≥ 6 mm. PPD is the depth from the free gingival margin to the base of the sulcus and it is measured in millimeters at several locations around the whole circumference of the tooth.
Percentages of sites PPDs ≥ 6 mm. | Change from baseline percentages of sites with PPDs ≥ 6 mm at six months
  Percentages of sites with PPDs ≥ 6 mm. PPD is the depth from the free gingival margin to the base of the sulcus and it is measured in millimeters at several locations around the whole circumference of the tooth.

SECONDARY OUTCOMES:
Operating time | Outcome measures will be recorded at baseline
  Time required to complete the procedure
Postoperative pain | Change from baseline pain at seven days
  Patient-related outcomes (pain) will be measured using visual analogue scale Minimum score 0 Maximum score 10 Higher score indicates worse outcome
Postoperative swelling | Change from baseline swelling at seven days
  Patient-related outcomes (swelling) will be measured using visual analogue scale Minimum score 0 Maximum score 10 Higher score indicates worse outcome
Postoperative bleeding | Change from baseline bleeding at seven days
  Patient-related outcomes (bleeding) will be measured using visual analogue scale Minimum score 0 Maximum score 10 Higher score indicates worse outcome
Postoperative bruising | Change from baseline bruising at seven days
  Patient-related outcomes (bruising) will be measured using visual analogue scale Minimum score 0 Maximum score 10 Higher score indicates worse outcome
Postoperative root sensitivity | Change from baseline root sensitivity at seven days
  Patient-related outcomes (root sensitivity) will be measured using visual analogue scale Minimum score 0 Maximum score 10 Higher score indicates worse outcome
Quality of life measures | Change from baseline GOHAI score at six months days
  Patient's quality of life will be evaluated using general oral health assessment index (GOHAI). The GOHAI has 12 negatively and positively worded items evaluating three dimensions of oral health related quality of life (physical function, pain or discomfort and psychosocial function).
  The score ranged from 0 to 60. The scores are maintained for the three items "able to swallow comfortably", able to eat without discomfort", "pleased with look of teeth", and reversed for the remaining nine items, so that a higher score was associated with a more positive oral health.

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Dental Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided